CLINICAL TRIAL: NCT01655199
Title: Measurement of Exertional Dyspnea in the Primary Care Setting in Patients With COPD, Phase III: Sensitivity of the Step Test to Detect Improvement in Dyspnea Following Bronchodilation in Patients With COPD
Brief Title: Sensitivity of the Step Test to Detect Improvement in Dyspnea Following Bronchodilation in Patients With Chronic Obstructive Pulmonary Disease
Acronym: CODEx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Benoit Borel, Postdoctoral fellow, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: CODEX-20819
Record Dates: First submitted 2012-07-25; First posted 2012-08-01 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Moderate Chronic Obstructive Pulmonary Disease; Severe Chronic Obstructive Pulmonary Disease; Dyspnea
Keywords: Chronic Obstructive Pulmonary Disease; Lung function; Exertional dyspnea; Exercise capacity; Pulmonary function; Pleural pressures
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Albuterol; Albuterol, Ipratropium Drug Combination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COPD group (Experimental): Moderate and/or severe COPD patients, corresponding to GOLD stages II and III.
  Interventions: Drug: Combination ipratropium/salbutamol or placebo (nebulization)

INTERVENTIONS:
Drug: Combination ipratropium/salbutamol or placebo (nebulization) — For the visit 2, COPD patients will be randomly assigned a combination of ipratropium/salbutamol or a placebo in a double-blind crossover design. For the visit 3, the other intervention drug will be assigned. The bronchodilation obtained with the medication will allow to determine if the 3-min step test is sensitive by detecting an improvement of exertional dyspnea following bronchodilation.
  Other Names: Combivent or placebo (nebulization)

SUMMARY:
During the previous phases of the project (Phase I and II), two new field tests have been designed and validated for an integration in a primary care setting in Chronic Obstructive Pulmonary Disease (COPD). These new field tests are 3-min paced-walk test (3MPWT) and 3-min paced step test (3MPST). If the validity and sensitivity of the TM3 could be highlighted, particularly by the reduction of dyspnea level following bronchodilatation, Phase II highlight that the 3MPST does not allow to detect this decrease of dyspnea after bronchodilatation. The use of too high step rates could explain these results through a hypothesis relative to neuromechanical coupling of dyspnea. The main objective of this trial is to follow the investigations on the sensitivity of 3MPST to detect the effects of pharmacological intervention on the exertional dyspnea in COPD patient. The hypothesis of this work is that the use of lower step rates cadences could allow to detect an improvement of exertional dyspnea following treatment-induced bronchodilatation, contrary to higher step rates.

DETAILED DESCRIPTION:
For this project, 40 patients with COPD will be recruited in 2 centres (in the Institute of Cardiology and Pneumology of Quebec and in the Chest Institute of Montreal). For each patient, three visits will be performed. During the first visit, baseline pulmonary function and maximal exercise capacity will be evaluated and the patients will be familiarized with step test proceedings. Between the different visits, a 3-7 days period will be respected. During the second and the third visits, 4 step tests will be performed at 4 different rates, following one of the two conditions (placebo or bronchodilatation). This project will propose two randomization levels. The first randomization will be relative to the choice of the condition used during the second visit (placebo ou bronchodilatation) and the second one for the rates order (14, 16, 20, 24 steps/min). During each performed exercise, cardiorespiratory and pulmonary parameters will be measured using a portable system.

ELIGIBILITY:
Inclusion Criteria:

* age higher than 50 years old
* smoking history ≥ 10 packs/year
* post-bronchodilator FEV1 between 30 and 80% of the predicted value and FEV1/FVC lesser than 70% as assessed in previous pulmonary function test (corresponding to GOLD stages II and III)

Exclusion Criteria:

* respiratory exacerbation within the preceding 6 weeks
* asthmatic condition
* significant O2 desaturation (SaO2 < 85%) at rest or during exercise
* presence of another pathology that could influence exercise tolerance or may prevent the realization of the step test
* subject having a pacemaker

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Symptom perception | change from baseline in Borg Scale at 3 min of exercise
  Patients will be asked to score their dyspnea and leg discomfort perception using a 10-point Borg scale.

SECONDARY OUTCOMES:
Cardiac and ventilatory outcomes | Change from baseline at 3 minutes of exercise
  Metabolic, cardiac and ventilatory parameters will be measured using a metabolic cart. Principal outcomes will be oxygen uptake (VO2), carbon dioxide output (VCO2), ventilation (VE), breathing frequency (BF), tidal volume (Vt) and heart rate (HR).
Inspiratory capacity | Change from baseline at the end of the exercise.
  Inspiratory capacity will be measured at rest and at the end of the 3-min step test (immediately following the assessment of dyspnea at 3 minutes).
Respiratory pressures and diaphragm EMG | Change from baseline at 1, 2 and 3 minutes of exercise
  Tidal excursion in pleural pressure will be measured using an oesophageal balloon-catheter system that will be positioned using standardized technique (n=40). Gastric and transdiaphragmatic pressures as well as the diaphragm electromyogram will be recorded in the 20 subjects studied at McGill University using a multipair esophageal electrode-balloon catheter.
Pulmonary function | At baseline and 60-min after the nebulization of either placebo and bronchodilator
  Pulmonary function will be measured by spirometry and plethysmography in the initial visit. In the subsequent visits, pulmonary function will be evaluated by spirometry before and 60-min after the nebulization of either placebo or bronchodilator.
Maximal oxygen consumption | Change from baseline at 1, 2 and 3 minutes of exercise
  Exercise capacity will be directly assessed following an incremental cycle exercise test. The exercise capacity was defined as the maximal oxygen consumption (VO2 peak, ml/kg/min) by direct measurements of gas exchanges.
Maximal inspiratory pressure (PImax) | Change from baseline after 3 minutes of exercise
  The maximum inspiratory pressure (PImax) will be measured during a sniff manoeuvre. These measurements will allow to construct the ratio of respiratory effort (tidal Pes/PImax) to thoracic displacement (VT/predicted VC), an index of neuromechanical coupling

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, M.D, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (2):
- Canada (2):
  - Montreal Chest Institute - McGill University, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec - Université Laval, Québec, Quebec